CLINICAL TRIAL: NCT03240276
Title: A Comparative Study of Sibling Oocytes, Which Examines Two Sperm Selection Methods for Top Quality of Spermatozoa , Prior Intracytoplasmic Sperm Injection (ICSI) Performance, and Their Effect on Embryo Quality and IVF Outcome: A Common Selection Method Based on Morphology (ICSI) vs. an Ultra Morphology Section Method - Intracytoplasmic Morphology Selected Sperm Injection (IMSI)
Brief Title: A Comparative Study of Sibling Oocytes: ICSI vs. the IMSI Sperm Selection Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-0070-17
Record Dates: First submitted 2017-07-31; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI Procedure (Active Comparator): The ICSI procedure is the standard procedure of selection and injection of sperm into the oocyte
  Interventions: Other: Standard ICSI procedure for sperm injection into oocyte
- IMSI Procedure (Active Comparator): The IMSI procedure is the injection of normal ultramorphological spermatozoa that have been selected using an inverted microscope with magnification of 6300x (MSOME)
  Interventions: Device: MSOME; Other: IMSI Procedure

INTERVENTIONS:
Other: Standard ICSI procedure for sperm injection into oocyte — The ICSI procedure is the standard procedure of selection and injection of sperm into oocytes
  Arms: ICSI Procedure
Device: MSOME — Selection of ultramorphologically normal spermatozoa using an inverted microscope with 6300x magnification
  Other Names: Motile Sperm Organelle Morphology Examination
  Arms: IMSI Procedure
Other: IMSI Procedure — Injection of sperm that has been selected by the MSOME method into oocytes
  Arms: IMSI Procedure

SUMMARY:
The aim of this research is to compare sibling oocytes using two sperm selection methods for choosing the best quality spermatozoa before they are injected into oocytes and the influence of each of these methods on embryo quality and IVF outcome.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-60
* Females aged 18-35
* Males defined as Moderate OTA or Isolated Teratozoospermia with less than 4% morphologically normal spermatozoa
* Patients with 0.5- 7% normal sperm according to MSOME analysis
* Females with normal FSH and AMH values
* Females who have retrieved at least 6 oocytes in previous cycles
* Couples who have had at least 2 failed IVF-ICSI cycles

Exclusion Criteria:

* Couples who have been exposed to heavy smoking, drugs and chronic diseases
* Males who have undergone testicular surgery (TESE) or defined as severe OTA
* Females with egg factor infertility

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of fertilization rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The fertilization rates of the ICSI and IMSI methods will be compared.
Comparison of embryo quality | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The embryo quality of the ICSI and IMSI methods will be compared.

SECONDARY OUTCOMES:
Implantation rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The implantation rates of the ICSI and IMSI methods will be compared.
Pregnancy rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The pregnancy rates of the ICSI and IMSI methods will be compared.
Miscarriage rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The miscarriage rates of the ICSI and IMSI methods will be compared.
Live birth rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The live birth rates of the ICSI and IMSI methods will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom Paz, MD, Principal Investigator — Hillel Yaffe Medical Center; Medeia Michaeli, PhD, Study Director — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No